CLINICAL TRIAL: NCT03915925
Title: Short-term Clinical Deterioration After Acute Pulmonary Embolism
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 1R01HS025979 (AHRQ)
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2019-07

CONDITIONS: Pulmonary Embolism
Keywords: right ventricle dysfunction; prediction model; functional outcomes
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, observational, multicenter cohort study to compare right ventricular dysfunction dependent and independent prognostic models for short-term serous adverse events in patients who are diagnosed with pulmonary embolism in the emergency department. Clinical endpoints are assessed at days 1-5. A thirty-day follow-up phone call is conducted to obtain further clinical endpoints and a quality of life assessment.

DETAILED DESCRIPTION:
The objective of this study is to compare right ventricular dysfunction (RVD)dependent and independent prognostic models for short-term serious adverse events in pulmonary embolism (PE) patients. The target population is emergency department (ED) patients with confirmed acute PE within 12 hours of ED presentation. The primary outcome is a composite of death, delayed circulatory or respiratory dysfunction, hypoxia, and reperfusion intervention within five days of PE diagnosis. Secondary outcomes will be nonfatal bleeding, recurrence of venous thromboembolism, and hypoxia requiring oxygen supplementation.

The specific aims are: 1) determine the incidence of death, circulatory and respiratory deterioration, and administration of reperfusion therapy within five days of PE; 2) determine functional outcomes 30 days after PE using the Pulmonary Embolism Quality of Life Questionnaire; 3) evaluate the sensitivity, specificity, and positive and negative likelihood ratios of each RVD assessment tool for clinical deterioration within five days of PE; and 4) derive a prediction model for clinical deterioration within five days of PE diagnosis.

Patients with confirmed PE will be assessed for hemodynamic stability at presentation, and then will be assessed for RVD. Normotensive PE patients without RVD will be assessed by a clinically derived model (sPESI or HESTIA) to determine if they are low risk or intermediate-low risk. The investigators will then determine incidence of the clinical endpoints during the subsequent 5 days, as well as 30 days later. The 30-day follow-up will also include administration of the validated Pulmonary Embolism Quality of Life questionnaire (PEmbQoL).

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18 years or older, with image confirmed acute pulmonary embolism diagnosed within 12 hours of ED presentation

Exclusion Criteria:

* Patients who decline any participation in the study
* Patients 17 years old and younger at the time of screening
* Radiologist's over read that determines that filling defects identified as acute emboli are instead either chronic, resolving, or unchanged after comparison to previous CT, if available
* If empiric anticoagulation or escalated intervention were initiated more than 12 hours before presentation to the recruiting ED
* Identification of either segmental or subsegmental intraluminal filling defects on CT that are considered to be clinically incidental and unrelated to primary diagnostic workup or ED presentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present to the emergency department with image confirmed acute pulmonary diagnosed within 12 hours of presentation
Sampling Method: Non-Probability Sample
Enrollment: 935 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Compare the risk ratio odds ratio of different PE risk stratification models for clinical Deterioration | Five days from diagnosis
  Provide and compare the number and proportion of patients with both composite and individual outcome of death, circulatory deterioration, respiratory deterioration, administration of reperfusion therapy

SECONDARY OUTCOMES:
Compare the prognostic accuracy of different right ventricular dysfunction parameters for predefined clinical deterioration outcomes within 5 days | 5 days from diagnosis
  Comparison of different Right Ventricular Dysfunction Assessments for Clinical deterioration within 5 days of PE diagnosis
Comparison of Patient Reported Pulmonary Embolism Functional outcomes at 30 days after Pulmonary Embolism Diagnosis | 30 days after PE diagnosis
  Comparison of functional outcomes between patients with and without Right ventricular dysfunction at presentation with higher scores indicating worse outcomes THe Pulmonary Embolism Quality of Life Questionnaire has six dimension of questions. Dimension scores are transformed into to scale from 0-100 with higher scores associated with worse outcomes.

OTHER OUTCOMES:
Development of prediction model for clinical deterioration outcomes within 5 days of PE presentation to emergency department | 5 days
  Use of logistic regression analysis to determine predictors of clinical deteriortion a=within 5 days of acute PE presentation at emergency department

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Weekes, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (6):
- United States (6):
  - San Diego Medical Center, San Diego, California
  - Christiana Care Health System, Newark, Delaware
  - Orlando Regional Medical Center, Orlando, Florida
  - Carolinas Medical Center - Main, Charlotte, North Carolina
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Univeristy of Utah Hospital, Salt Lake City, Utah